CLINICAL TRIAL: NCT03103009
Title: Treatment Plan for an Individual Patient With Pasireotide for Hyperinsulinemic Hypoglycemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0393
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Hyperinsulinemic Hypoglycemia; Post Gastrointestinal Tract Surgery Hypoglycaemia
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — pasireotide

STUDY DESIGN:
Intervention Model Description: Treatment Plan for an individual patient with pasireotide for Hyperinsulinemic Hypoglycemia (Compassionate Use Protocol for Pasireotide)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- pasireotide (Experimental): Interventions - One patient will be given a drug, pasireotide (Signifor), on a compassionate use basis for treatment of post-gastric bypass hypoglycemia. The minimal dose will be 0.3 mg subcutaneous daily and the maximal dose will be 0.6 mg subcutaneous twice daily. The patient may continue treatment with pasireotide indefinitely unless the patient experiences unacceptable toxicity, disease progression and/or treatment is discontinued at the discretion of the treating physician or Novartis or withdrawal of consent.
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide — Somatostatin analogues are a last resort for medical intervention in hyperinsulinemic hypoglycemia (HH). The hypoglycemia is very debilitating and can be even life threatening. There is limited experience with pasireotide in hyperinsulinemic hypoglycemia (only one publication); there is more experience with octreotide, both in adults and children and successful interventions with octreotide in hyperinsulinemic hypoglycemia have been published. Pasireotide via its different somatostatin receptor binding profile has clear effects on insulin, glucagon and incretin secretion and can ultimately lead to hyperglycemia. This mode of action (especially the effects on insulin and incretin secretion) could be very useful in the setting of hyperinsulinemic hypoglycemia.
  Other Names: Signifor

SUMMARY:
Somatostatin analogues are a last resort for medical intervention in hyperinsulinemic hypoglycemia (HH). The hypoglycemia is very debilitating and can be even life threatening. There is limited experience with pasireotide in hyperinsulinemic hypoglycemia (only one publication); there is more experience with octreotide, both in adults and children successful interventions with octreotide in hyperinsulinemic hypoglycemia have been published. Pasireotide via its different somatostatin receptor binding profile has clear effects on insulin, glucagon and incretin secretion and can ultimately lead to hyperglycemia. This mode of action (especially the effects on insulin and incretin secretion) could be very useful in the setting of hyperinsulinemic hypoglycemia.

DETAILED DESCRIPTION:
Hyperinsulinemic hypoglycemia as a complication of gastric bypass surgery has been reported to occur between 6 months to 8-10 years after gastric bypass surgery. Although reported as a rare complication from surgery, the incidence is likely higher due to the condition being missed in many patients or being misdiagnosed as dumping syndrome. Unlike dumping syndrome which often presents early in the post-operative course and improves with dietary modification, patients with hyperinsulinemic hypoglycemia have severe postprandial hypoglycemia and sometimes fasting hypoglycemia with symptoms worsening over time despite dietary modification. Calcium stimulation testing often localizes the area of the pancreas where hyperinsulinemia is occurring due to islet cell dysfunction. The pathophysiology of islet cell hypertrophy with Nesidioblastosis is poorly understood. One theory is an increase in glucagon-like peptide-1 (GLP-1) concentration may be responsible for islet cell expansion and subsequent hyperinsulinemic hypoglycemia.

Unfortunately, hyperinsulinemia hypoglycemia is incapacitating where patients are restricted from driving, are unable to work, and must always have someone present with glucagon due to the acute severe onset of neuroglycopenia. Surgery to resect the area of the pancreas with Nesidioblastosis has a low success rate of about 60% with many patients developing type 1 diabetes as a result of pancreatic resection. Medical treatment options include calcium channel blockers, Diazoxide, and Octreotide yet patients often fail these treatments as well. Pasireotide would likely be a better option than the current medical therapy available. With Pasireotide, the inhibition of insulin release through inhibiting the somatostatin receptors as well as possible GLP-1 inhibition causing hyperglycemia should reduce hypoglycemic episodes in these patients.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

1. Male or female patients aged 18 years or older
2. Patients with a confirmed diagnosis of hyperinsulinemic hypoglycemia, if possible by genetic testing
3. Patients not controlled by medical therapies (e.g. diazoxide or octreotide) and/or pancreatic surgery or patients not eligible for surgery
4. WHO/ ECOG Performance Status of 0-2.
5. Life expectancy ≥12 weeks
6. Adequate end organ function as defined by:

   No evidence of significant liver disease:
   * Serum total bilirubin ≤1.5 x ULN
   * INR < 1.3
   * ALT and AST ≤ 2 x ULN,
   * Alkaline phosphatase ≤ 2.5 x ULN
7. Written informed consent obtained prior to treatment to be consistent with local regulatory requirements
8. Is suffering from a serious or life-threatening disease or condition
9. Does not have access to a comparable or satisfactory alternative treatment (i.e., comparable or satisfactory treatment is not available or does not exist)
10. Is not eligible for participation in any of the IMP's ongoing clinical trials or has recently completed a clinical trial that has been terminated and, after considering other options (e.g., trial extensions, amendments, etc.), the clinical team has determined that treatment is necessary and there are no other feasible alternatives for the patient
11. There are meaningful human clinical data to support an assessment that the potential benefits to patient outweigh risks.
12. Meets any other relevant medical criteria for compassionate use of the investigational product
13. Is not being transferred from an ongoing clinical trial for which they are still eligible

Exclusion Criteria:

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. Patients with a known hypersensitivity to somatostatin analogs or any component of the pasireotide LAR or s.c. formulations.
2. Patients with abnormal coagulation (PT or aPTT elevated by 30% above normal limits).
3. Patients on continuous anticoagulation therapy. Patients who were on anticoagulant therapy must complete a washout period of at least 10 days and have confirmed normal coagulation parameters before study inclusion.
4. Patients currently using warfarin / warfarin derivatives
5. Patients with symptomatic cholelithiasis.
6. Patients who are not biochemically euthyroid. Patients with known history of hypothyroidism are eligible if they are on adequate and stable replacement thyroid hormone therapy for at least 3 months.
7. QT-related exclusion criteria: :

   * QTcF at screening > 450 msec in males and QTcF > 460 msec
   * History of syncope or family history of idiopathic sudden death
   * Sustained or clinically significant cardiac arrhythmias
   * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
   * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
   * Family history of long QT syndrome
   * Concomitant medications known to prolong the QT interval.
   * Potassium < or = 3.5 mmol/L
8. Patients who have any severe and/or uncontrolled medical conditions :

   * Uncontrolled diabetes as defined by HbA1c > 8%,
   * Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunodeficiency, including a positive HIV test result (ELISA and Western blot). An HIV test will not be required; however, previous medical history will be reviewed.
   * Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with this study treatment.
   * Life-threatening autoimmune and ischemic disorders.
9. Patients who have a history of another primary malignancy, with the exception of locally excised non-melanoma skin cancer and carcinoma in situ of uterine cervix. Patients who have had no evidence of disease from another primary cancer for 1 or more years are allowed to participate in the study.
10. Patients with history of liver disease, such as cirrhosis or chronic active hepatitis B or C
11. Presence of Hepatitis B surface antigen (HbsAg)
12. Presence of Hepatitis C antibody (anti-HCV)
13. History of, or current alcohol misuse/abuse within the past 12 months.
14. Known gallbladder or bile duct disease, acute or chronic pancreatitis
15. Patients with hypomagnesaemia (< 0.7 mmol/L)
16. Patients with a history of non-compliance to medical regimens or who are considered potentially
17. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
    * Combination of any two of the following (a+b or a+c, or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
18. If the patient is a sexually active male he is excluded unless he agrees to use a condom during intercourse while taking pasireotide and for 3 months after stopping pasireotide medication . They should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Recording of Hypoglycemic events | Up to 2 years
  The primary outcome is the number of hypoglycemic events occurring.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lawler, MD, Principal Investigator — University of Colorado, Denver; Mike McDermott, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with Novartis.